CLINICAL TRIAL: NCT04591457
Title: The Efficacy, Safety, and Immunogenicity Study Comparing an Insulin Glargine Biosimilar Sansulin® Log-G With Its Reference Lantus® in Patients With Type 2 Diabetes Mellitus
Brief Title: The Efficacy, Safety, and Immunogenicity Study Comparing an Insulin Glargine Biosimilar Sansulin Log-G to Lantus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr Tri Juli Edi Tarigan, SpPD-KEMD, Endocrinologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaU-03
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Insulin glargine biosimilar; diabetes mellitus; efficacy; safety; immunogenicity
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Glargine Sansulin (Experimental): Drug product Insulin Glargine, Sansulin Log-G 100 IU/mL (PT. Sanbe Farma)
  Interventions: Drug: Insulin Glargine Sansulin
- Insulin Glargine Lantus (Active Comparator): Drug product Insulin Glargine, Pen Injector [Lantus] 100 IU/mL (PT. Sanofi-Aventis)
  Interventions: Drug: Insulin Glargine Pen Injector [Lantus]

INTERVENTIONS:
Drug: Insulin Glargine Sansulin — Insulin Glargine (Sansulin Log-G) once daily at individually adjusted dose
  Other Names: Sansulin
  Arms: Insulin Glargine Sansulin
Drug: Insulin Glargine Pen Injector [Lantus] — Insulin Glargine (Lantus) once daily at individually adjusted dose
  Other Names: Lantus
  Arms: Insulin Glargine Lantus

SUMMARY:
This is an open-label randomised multicenter clinical study to investigate efficacy, safety, and immunogenicity of the drug products: Insulin Glargine biosimilar ® Log-G and its reference Lantus® in type 2 diabetes mellitus patients

DETAILED DESCRIPTION:
Sansulin® Log-G is an insulin glargine biosimilar. For a biosimilar, its efficacy, safety, and immunogenicity should be compared head-to-head with its reference product in at least non-inferiority study. Immunogenicity assessment should always be done because it is influenced by so many factors, from nature of the drug substance until patient and disease related factors. Moreover its consequences also vary considerably, from clinically irrelevant to serious and life-threatening. Immunogenicity of a biosimilar should always be investigated in humans, since animal data are usually not predictive of the immune response in humans.

Since blinding of study participants is likely unfeasible, at least anti-drug antibodies should be determined in a blinded fashion. Since anti-insulin antibodies develop early, then 6 months duration of study is adequate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DM type 2, age at least 18 years, both genders.
2. T2DM patients who have been diagnosed for > 1 year, and have been treated with one oral antidiabetic at stable doses for > 3 months prior to screening, have BMI of 18.0 to 35.0 kg/m2 inclusive, and HbA1C of > 7.0% and insulin-naive.
3. Patients who are cooperative, reliable, and agree to have regular injections of insulin, and are willing to comply with protocol procedure (willing to sign the informed consent).
4. Female patients with adequate protection from conception. Females of childbearing potential must use a reliable method of birth control during the study (barrier-method or IUD). Women with history of bilateral tubal ligation, or with total hysterectomy, or who are 2 years postmenopausal are also eligible.

Exclusion Criteria:

1. Pregnancy (confirmed by a positive urine pregnancy test) or lactation.
2. History of severe hypoglycemia during the last year (blood glucose level <50 mg/dl with transient dysfunction of central nervous system without other apparent cause)
3. History of diabetic ketoacidosis > 2x within the last year.
4. Having hyperglycemia hyperosmolar status (HHS)
5. Renal impairment (eGFR < 30 mL/min).
6. An employee of the Investigator or the Sponsor.
7. Participating in another clinical study within the past 3 months.
8. Receiving any immunosuppressants, including corticosteroids or cytostatics within the last year or during the study.
9. Receiving any drug or supplement with hypoglycemic activity (except oral antidiabetics) within 4 weeks prior to screening and during the study.
10. Receiving any drug with hyperglycemic activity within 4 weeks prior to screening and during the study (eg. second generation antipsychotics, corticosteroids, tacrolimus, protease inhibitors).
11. Have undergone pancreatectomy or pancreas / islet cell transplant.
12. Mental disorder
13. Any malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 24 weeks
  Change in HbA1c level after 24 weeks of therapy compared to baseline value
Number of patients | 24 weeks
  Number of patients with HbA1c < 7%
Anti-insulin antibodies (AIAs) | 24 weeks
  Change in anti-insulin antibodies (AIAs) after 24 weeks of therapy compared to baseline value

SECONDARY OUTCOMES:
FBG & PPBG | 24 weeks
  Change in FBG & PPBG compared to baseline
Hypoglycemia | 24 weeks
  Incidence and severity of hypoglycemia
Weight gain | 24 weeks
  Incidence of weight gain
Adverse events | 24 weeks
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tri Juli Edi Tarigan, Principal Investigator — Cipto Mangunkusumo General Hospital/Faculty of Medicine Universitas Indonesia
Locations (1):
- Department of Internal Medicine Cipto Mangunkusumo General Hospital, Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knezevic I. Evaluation of similar biotherapeutic products (SBPs): scientific principles and their implementation. Biologicals. 2011 Sep;39(5):256-61. doi: 10.1016/j.biologicals.2011.08.008. Epub 2011 Sep 9. PMID 21907589